CLINICAL TRIAL: NCT07226635
Title: Pharmacokinetic Interaction Trial of Clofutriben With Midazolam and Prednisolone
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPI-62-CL-1004
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: midazolam (Experimental): Drug: 2 single oral doses of midazolam
  Interventions: Drug: midazolam
- 2 single oral doses of prednisolone (Experimental): 2 single oral doses of prednisolone
  Interventions: Drug: 2 single oral doses of prednisolone
- clofutriben once daily for 16 days (Experimental): clofutriben once daily for 16 days
  Interventions: Drug: clofutriben once daily for 16 days

INTERVENTIONS:
Drug: midazolam — Drug: 2 single oral doses of midazolam ,
  Arms: Experimental: midazolam
Drug: clofutriben once daily for 16 days — clofutriben once daily for 16 days
  Arms: clofutriben once daily for 16 days
Drug: 2 single oral doses of prednisolone — 2 single oral doses of prednisolone
  Arms: 2 single oral doses of prednisolone

SUMMARY:
Drug: 2 single oral doses of midazolam, 2 single oral doses of prednisolone , and clofutriben once daily for 16 days.

DETAILED DESCRIPTION:
Approximately 16 healthy male and female participants will be enrolled at a single center in the US. Each participant will receive 2 single oral doses of midazolam , 2 single oral doses of prednisolone, and clofutriben once daily for 16 days. On each day that midazolam is administered, blood samples for midazolam analysis in plasma will be collected for 24 hours. On each day that prednisolone is administered, blood samples for prednisolone, prednisone, and 6β-hydroxyprednisolone analyses in plasma will be collected for 24 hours.

Blood samples for clofutriben and metabolite (AS2570469) analyses in plasma will be collected for 24 hours after the first dose and during 2 intervals at steady state. Blood samples for cortisol and cortisone analyses will be collected for 24 hours after administration of prednisolone, clofutriben, and both trial interventions together, and prior to dosing of either trial intervention. Urine will be collected for analysis of clofutriben, prednisolone, and metabolites. Feces will be collected for analysis of clofutriben and metabolites. Safety and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 75 years of age,
* Body mass index of 18 to 35 kg/m2,
* Taking no medications,
* Are considered by the investigator to be in good general health.

Exclusion Criteria:

* In the opinion of the investigator, the participant is not suitable for entry into the trial or has any contraindication to midazolam or prednisolone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-10-03 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam. | 24 hours from dose
  It will be concluded that there is no relevant interaction of clofutriben on midazolam if the 90% CIs for the Cmax ratios (midazolam + clofutriben)/midazolam alone) are contained within the [80%, 125%] interval.
AUC0-t of midazolam | 24 hours from dose
  : It will be concluded that there is no relevant interaction of clofutriben on midazolam if the 90% CIs for the AUC0-t (midazolam + clofutriben)/midazolam alone) are contained within the [80%, 125%] interval.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided